CLINICAL TRIAL: NCT02989454
Title: Persistent Symptoms and Early Incomplete Recovery After Acute Stress-induced Cardiomyopathy: Is There Ongoing Heart Distress? The HEROIC Study
Acronym: HEROIC
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2/005/15
Record Dates: First submitted 2016-03-24; First posted 2016-12-12 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Tako-tsubo Cardiomyopathy
MeSH Terms: conditions — Takotsubo Cardiomyopathy | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Samples for genetic analysis will be stored.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tako Tsubo Cardiomyopathy patients: Any patient who has suffered from Tako Tsubo Cardiomyopathy since 2011.
  Interventions: Other: Assessment of exercise capacity and cardiac energetics

INTERVENTIONS:
Other: Assessment of exercise capacity and cardiac energetics — Cardiopulmonary exercise testing and Magnetic Resonance Spectroscopy
  Other Names: MRI, MRS and CPEX

SUMMARY:
Acute stress induced (Tako-tsubo) cardiomyopathy (TTC) or broken heart syndrome, a condition typically occurring after acute stress has a death rate similar to heart attacks and is frequently associated with long-term symptoms (fatigue and exercise limitation). There are no effective therapies. The investigators have recently showed that there is a profound shortage of energy in the hearts of Tako Tsubo Cardiomyopathy patients in the days after acute presentation with only partial recovery by four months. The investigators would now like to establish whether this recovers after at least one year, or persists, and also to investigate the mechanisms responsible for exercise limitation after recovery from the acute phase.

DETAILED DESCRIPTION:
Tako Tsubo Cardiomyopathy presents with sudden onset of chest pain that mimics a myocardial infarction (MI) and is precipitated by major emotional/physical stress. Classically, the coronary arteries are normal and yet, the left ventricular (LV) angiogram shows a characteristic, extensive and severe wall motion abnormality, some develop cardiogenic shock, cardiac rupture or embolic stroke. In the weeks following onset, the wall motion abnormalities gradually recover: this led to the assumption that Tako Tsubo Cardiomyopathy is self-limiting, reinforced by the absence of myocardial damage on cardiac Magnetic Resonance Imaging. However, the investigators and others have shown that Tako Tsubo Cardiomyopathy recovery is not rapid, being characterised by severe global oedema, which persists for 3-4 months after presentation. The investigators showed profound decrease in cardiac energetics during the acute Tako Tsubo Cardiomyopathy phase compared to healthy controls. This improved significantly at follow up but remained reduced compared to healthy controls.

These objective findings of incompletely resolved myocardial oedema and energetic impairment are in contrast with the more rapid apparent recovery of Left Ventricular Ejection Fraction but are in keeping with the persistence of symptoms previously reported in literature and with the investigators' own clinical observations from the Tako Tsubo Cardiomyopathy follow-up clinic at the institution.

The persistence of symptoms (fatigue, recurrent chest pains, decreased exercise capacity) could be due to either:

1. Subclinical degree of impairment in cardiac energetics/function (reflecting either an even more prolonged status of incomplete recovery or a pre-existent cardiomyopathy) which despite a normalised for almost normalised ejection fraction at rest results in cardiac limitation during exercise, or
2. Physical deconditioning after an acute, severe illness.

ELIGIBILITY:
Inclusion Criteria:

* Any patient diagnosed with Tako Tsubo Cardiomyopathy in Aberdeen, Glasgow and Inverness since 2011.

Exclusion Criteria:

* Contraindication to magnetic resonance scanning such as an implantable cardiac device, etc for those undergoing magnetic resonance imaging only (they can attend for cardiopulmonary exercise testing and bloods).
* Inability to exercise on a treadmill (they can attend for magnetic resonance imaging and bloods).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient that has been diagnosed with Tako Tsubo Cardiomyopathy since 2011.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-08; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Cardiac energetics by cardiac magnetic resonance imaging | One year or longer after diagnosis
  Cardiac magnetic resonance imaging and spectroscopy

SECONDARY OUTCOMES:
Exercise capacity | One year or longer after diagnosis
  Cardiopulmonary exercise testing

CONTACTS AND LOCATIONS:
Overall Officials: Dana Dawson, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- Cardiac Research Office, Aberdeen Royal Infirmary, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prasad A, Lerman A, Rihal CS. Apical ballooning syndrome (Tako-Tsubo or stress cardiomyopathy): a mimic of acute myocardial infarction. Am Heart J. 2008 Mar;155(3):408-17. doi: 10.1016/j.ahj.2007.11.008. Epub 2008 Jan 31. PMID 18294473
- [Background] Sy F, Basraon J, Zheng H, Singh M, Richina J, Ambrose JA. Frequency of Takotsubo cardiomyopathy in postmenopausal women presenting with an acute coronary syndrome. Am J Cardiol. 2013 Aug 15;112(4):479-82. doi: 10.1016/j.amjcard.2013.04.010. Epub 2013 May 16. PMID 23683950
- [Background] Sharkey SW, Windenburg DC, Lesser JR, Maron MS, Hauser RG, Lesser JN, Haas TS, Hodges JS, Maron BJ. Natural history and expansive clinical profile of stress (tako-tsubo) cardiomyopathy. J Am Coll Cardiol. 2010 Jan 26;55(4):333-41. doi: 10.1016/j.jacc.2009.08.057. PMID 20117439
- [Background] Elesber AA, Prasad A, Lennon RJ, Wright RS, Lerman A, Rihal CS. Four-year recurrence rate and prognosis of the apical ballooning syndrome. J Am Coll Cardiol. 2007 Jul 31;50(5):448-52. doi: 10.1016/j.jacc.2007.03.050. Epub 2007 Jul 16. PMID 17662398
- [Background] Eitel I, von Knobelsdorff-Brenkenhoff F, Bernhardt P, Carbone I, Muellerleile K, Aldrovandi A, Francone M, Desch S, Gutberlet M, Strohm O, Schuler G, Schulz-Menger J, Thiele H, Friedrich MG. Clinical characteristics and cardiovascular magnetic resonance findings in stress (takotsubo) cardiomyopathy. JAMA. 2011 Jul 20;306(3):277-86. doi: 10.1001/jama.2011.992. PMID 21771988
- [Background] Neil C, Nguyen TH, Kucia A, Crouch B, Sverdlov A, Chirkov Y, Mahadavan G, Selvanayagam J, Dawson D, Beltrame J, Zeitz C, Unger S, Redpath T, Frenneaux M, Horowitz J. Slowly resolving global myocardial inflammation/oedema in Tako-Tsubo cardiomyopathy: evidence from T2-weighted cardiac MRI. Heart. 2012 Sep;98(17):1278-84. doi: 10.1136/heartjnl-2011-301481. Epub 2012 Jul 11. PMID 22791656
- [Background] Horowitz JD, Nguyen TH. Role of echocardiography in tako-tsubo cardiomyopathy: beyond diagnosis? JACC Cardiovasc Imaging. 2014 Feb;7(2):130-2. doi: 10.1016/j.jcmg.2013.09.021. No abstract available. PMID 24524742
- [Background] Singh K, Carson K, Usmani Z, Sawhney G, Shah R, Horowitz J. Systematic review and meta-analysis of incidence and correlates of recurrence of takotsubo cardiomyopathy. Int J Cardiol. 2014 Jul 1;174(3):696-701. doi: 10.1016/j.ijcard.2014.04.221. Epub 2014 Apr 26. PMID 24809923
- [Background] Chen X, Lee G, Maher BS, Fanous AH, Chen J, Zhao Z, Guo A, van den Oord E, Sullivan PF, Shi J, Levinson DF, Gejman PV, Sanders A, Duan J, Owen MJ, Craddock NJ, O'Donovan MC, Blackman J, Lewis D, Kirov GK, Qin W, Schwab S, Wildenauer D, Chowdari K, Nimgaonkar V, Straub RE, Weinberger DR, O'Neill FA, Walsh D, Bronstein M, Darvasi A, Lencz T, Malhotra AK, Rujescu D, Giegling I, Werge T, Hansen T, Ingason A, Noethen MM, Rietschel M, Cichon S, Djurovic S, Andreassen OA, Cantor RM, Ophoff R, Corvin A, Morris DW, Gill M, Pato CN, Pato MT, Macedo A, Gurling HM, McQuillin A, Pimm J, Hultman C, Lichtenstein P, Sklar P, Purcell SM, Scolnick E, St Clair D, Blackwood DH, Kendler KS; GROUP investigators; International Schizophrenia Consortium. GWA study data mining and independent replication identify cardiomyopathy-associated 5 (CMYA5) as a risk gene for schizophrenia. Mol Psychiatry. 2011 Nov;16(11):1117-29. doi: 10.1038/mp.2010.96. Epub 2010 Sep 14. PMID 20838396
- [Background] Ashbrook DG, Williams RW, Lu L, Hager R. A cross-species genetic analysis identifies candidate genes for mouse anxiety and human bipolar disorder. Front Behav Neurosci. 2015 Jul 1;9:171. doi: 10.3389/fnbeh.2015.00171. eCollection 2015. PMID 26190982
- [Background] McCalmon SA, Desjardins DM, Ahmad S, Davidoff KS, Snyder CM, Sato K, Ohashi K, Kielbasa OM, Mathew M, Ewen EP, Walsh K, Gavras H, Naya FJ. Modulation of angiotensin II-mediated cardiac remodeling by the MEF2A target gene Xirp2. Circ Res. 2010 Mar 19;106(5):952-60. doi: 10.1161/CIRCRESAHA.109.209007. Epub 2010 Jan 21. PMID 20093629
- [Background] Pison L, De Vusser P, Mullens W. Apical ballooning in relatives. Heart. 2004 Dec;90(12):e67. doi: 10.1136/hrt.2004.046813. PMID 15547001
- [Background] Kumar G, Holmes DR Jr, Prasad A. "Familial" apical ballooning syndrome (Takotsubo cardiomyopathy). Int J Cardiol. 2010 Oct 29;144(3):444-5. doi: 10.1016/j.ijcard.2009.03.078. Epub 2009 Apr 17. PMID 19375184
- [Background] Sharkey SW, Lips DL, Pink VR, Maron BJ. Daughter-mother tako-tsubo cardiomyopathy. Am J Cardiol. 2013 Jul 1;112(1):137-8. doi: 10.1016/j.amjcard.2013.02.063. Epub 2013 Apr 2. PMID 23561588
- [Background] Caretta G, Robba D, Vizzardi E, Bonadei I, Raddino R, Metra M. Tako-tsubo cardiomyopathy in two sisters: a chance finding or familial predisposition? Clin Res Cardiol. 2015 Jul;104(7):614-6. doi: 10.1007/s00392-015-0837-0. Epub 2015 Mar 6. No abstract available. PMID 25743177
- [Derived] Khan H, Rudd A, Gamble DT, Mezincescu AM, Cheyne L, Horgan G, Dhaun N, Newby DE, Dawson DK. Renin-Angiotensin and Endothelin Systems in Patients Post-Takotsubo Cardiomyopathy. J Am Heart Assoc. 2022 Jul 19;11(14):e025989. doi: 10.1161/JAHA.122.025989. Epub 2022 Jul 13. PMID 35861811
- [Derived] Scally C, Rudd A, Mezincescu A, Wilson H, Srivanasan J, Horgan G, Broadhurst P, Newby DE, Henning A, Dawson DK. Persistent Long-Term Structural, Functional, and Metabolic Changes After Stress-Induced (Takotsubo) Cardiomyopathy. Circulation. 2018 Mar 6;137(10):1039-1048. doi: 10.1161/CIRCULATIONAHA.117.031841. Epub 2017 Nov 11. PMID 29128863